CLINICAL TRIAL: NCT00532844
Title: A Phase 2 Randomized Open-label 2-Treatment 2-Sequence 2-Period Crossover PK Study to Compare Plasma Concentrations of BH4 in Subjects With Endothelial Dysfunction Following 14 Days of Treatment by 2 Regimens: 6R-BH4 With Vitamin C and 6R-BH4 Alone
Brief Title: A Phase 2, Pharmacokinetic (PK) Study of 6R-BH4 Alone or 6R-BH4 With Vitamin C in Subjects With Endothelial Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HTN-002
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Results first posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-04

CONDITIONS: Endothelial Dysfunction
Keywords: 6R-BH4; BH4; BH4 deficiency; sapropterin dihydrochloride; endothelial dysfunction; NO; Hypertension; Nitric Oxide; Vitamin C
MeSH Terms: conditions — Phenylketonurias; Hypertension | interventions — sapropterin; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sapropterin dihydrochloride (Experimental): Sapropterin dihydrochloride 5 mg/kg twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14 and Day 28.
  Interventions: Drug: Sapropterin Dihydrochloride
- Sapropterin dihydrochloride+Vitamin C (Experimental): Sapropterin dihydrochloride 5 mg/kg and 500 mg Vitamin C twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14 and Day 28.
  Interventions: Drug: Sapropterin Dihydrochloride and Vitamin C

INTERVENTIONS:
Drug: Sapropterin Dihydrochloride — Sapropterin Dihydrochloride 5 mg/kg twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14 and Day 28.
  Other Names: 6R-BH4
  Arms: Sapropterin dihydrochloride
Drug: Sapropterin Dihydrochloride and Vitamin C — Sapropterin Dihydrochloride 5 mg/kg and 500 mg Vitamin C twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14 and Day 28.
  Other Names: 6R-BH4 and Vitamin C
  Arms: Sapropterin dihydrochloride+Vitamin C

SUMMARY:
This Phase 2, randomized, open-label, 2-treatment, 2-sequence, 2-period crossover, pharmacokinetic (PK) study will compare plasma concentrations of BH4 in subjects with endothelial dysfunction following 14 days of treatment by each of 2 regimens: sapropterin dihydrochloride with vitamin C and sapropterin dihydrochloride alone.

DETAILED DESCRIPTION:
This was a Phase 2, randomized, open-label, 2-treatment, 2-sequence, 2-period crossover, pharmacokinetic (PK) study designed to compare the plasma concentrations of BH4 in subjects with endothelial dysfunction following 14 days of treatment by each of 2 regimens: sapropterin dihydrochloride with vitamin C and sapropterin dihydrochloride alone. Each subject received each regimen; the 2 treatment groups varied only in the sequence of the 2 regimens. The washout period between treatment regimens comprised the 1 day period between the last dose of study drug under the first regimen and the first dose of study drug under the second regimen (Day 14 morning to Day 15 morning).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures.
* Age is ≥ 18 years and ≤ 75 years.
* Willing and able to comply with all study procedures.
* If currently receiving treatment with or taking any of the following supplements, be willing and able to discontinue taking them throughout the treatment period:

  * Vit C supplements
  * Multivitamins containing vit C
  * Any other dietary supplements, nutraceuticals, or other over- the-counter products containing vit C
  * Vitamin E-containing supplements
* History of cardiovascular disease or cardiovascular risk factors, eg, stable and well-controlled Type 2 diabetes, peripheral arterial disease, obesity, smoking, hypercholesterolemia
* Endothelial dysfunction, documented at screening by an abnormal peripheral arterial tonometry (PAT) of ≤ 1.70.
* Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
* Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to screening, or who have had total hysterectomy.

Exclusion Criteria:

* Hypertension secondary to other medical conditions (e.g., renal failure or steroid usage).
* Concurrent disease or condition that would interfere with study participation or safety, such as bleeding disorders; history of syncope or vertigo; severe gastroesophageal reflux disease (GERD); heart failure; symptomatic coronary disease; arrhythmia; serious neurologic disorders, including seizures; organ transplant; or organ failure.
* Type 2 diabetics that are uncontrolled, unstable, newly diagnosed, or have changed therapy in the last three months and all Type 1 diabetics.
* Any severe comorbid condition that would limit life expectancy to < 6 months.
* Serum creatinine > 2.0 mg/dL, or hepatic enzyme concentrations > 2 times the upper limit of normal
* HIV infection, hepatic cirrhosis, other preexisting liver disease, or positive HIV, Hepatitis B or C test at screening.
* Concomitant treatment with:

  * Drugs known to inhibit folate metabolism (e.g., methotrexate)
  * Levodopa
  * A phosphodiesterase (PDE) 5 inhibitor (e.g., Viagra®, Cialis®, Levitra®, or Revatio®)
  * A PDE 3 inhibitor (e.g., cilostazol, milrinone, or vesnarinone)
* Use of any investigational product or investigational medical device within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Myocardial infarction, stroke, or surgery within the last 60 days prior to screening.
* History of alcohol and/or drug abuse or a positive alcohol or drug test at screening.
* Previous treatment with any formulation of BH4.
* Has known hypersensitivity to 6R-BH4 or its excipients.
* Pregnant or breastfeeding at screening, or planning to become pregnant (self or partner) at any time during the study.
* Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Nwose, MD, Study Director — BioMarin Pharmaceutical
Locations (1):
- Hackensack, New Jersey, United States

REFERENCES:
- See also: BioMarin Pharmaceutical Inc. website — http://www.bmrn.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-center study.
Pre-assignment Details: A total of 52 subjects were randomized into the study and received study drug.
  Of these, 4 subjects were enrolled under an earlier version of the protocol that used different eligibility criteria and were monitored according to different data collection procedures.
  Only the 48 subjects enrolled under the final protocol were included in the analyses.
Groups:
- Sapropterin Dihydrochloride 10mg/kg First; Then Sapropterin Dihydrochloride 10mg/kg and Vitamin C: Sequence A: Sapropterin dihydrochloride as the first treatment followed by sapropterin dihydrochloride and vitamin C
  Treatment Regimen 1: Sapropterin dihydrochloride 5 mg/kg twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14.
  Treatment Regimen 2: Sapropterin dihydrochloride 5 mg/kg + 500 mg vitamin C twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 28
  The washout period of 1 day comprised between treatment regimens.
- Sapropterin Dihydrochloride 10mg/kg and Vitamin C First; Then Sapropterin Dihydrochloride 10mg/kg: Sequence B: Sapropterin dihydrochloride and vitamin C as the first treatment followed by sapropterin dihydrochloride.
  Treatment Regimen 2: Sapropterin dihydrochloride 5 mg/kg + 500 mg vitamin C twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14.
  Treatment Regimen 1: Sapropterin dihydrochloride 5 mg/kg twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal Day 28.
  The washout period of 1 day comprised between treatment regimens.
Period: Treatment Period - Day 1 to Day 14
Arm/Group | Sapropterin Dihydrochloride 10mg/kg First; Then Sapropterin Dihydrochloride 10mg/kg and Vitamin C | Sapropterin Dihydrochloride 10mg/kg and Vitamin C First; Then Sapropterin Dihydrochloride 10mg/kg
Started | 24 (Only the 48 subjects enrolled in the final protocol are included in the participant flow.) | 24 (Only the 48 subjects enrolled in the final protocol are included in the participant flow.)
Completed | 24 | 23
Not Completed | 0 | 1
Not completed — Withdrawal of consent | 0 | 1
Period: Washout (1 Day)
Arm/Group | Sapropterin Dihydrochloride 10mg/kg First; Then Sapropterin Dihydrochloride 10mg/kg and Vitamin C | Sapropterin Dihydrochloride 10mg/kg and Vitamin C First; Then Sapropterin Dihydrochloride 10mg/kg
Started | 24 | 23
Completed | 24 | 23
Not Completed | 0 | 0
Period: Treatment Period - Day 15 to Day 28
Arm/Group | Sapropterin Dihydrochloride 10mg/kg First; Then Sapropterin Dihydrochloride 10mg/kg and Vitamin C | Sapropterin Dihydrochloride 10mg/kg and Vitamin C First; Then Sapropterin Dihydrochloride 10mg/kg
Started | 24 | 23
Completed | 20 | 23
Not Completed | 4 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Personal reasons | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — withdrawal of consent | 1 | 0

BASELINE CHARACTERISTICS:
Population: Four subjects, were enrolled prior to change in the study design from a parallel to a crossover study. These four subjects were not included in the baseline analysis population as they only received one treatment (either sapropterin dihydrochloride alone or sapropterin dihydrochloride and vitamin C) for the full 29-day duration of the study.
Groups:
- Sapropterin Dihydrochloride 10mg/kg First, Then Sapropterin Dihydrochloride 10mg/kg and Vitamin C: Sequence A: Sapropterin dihydrochloride as the first treatment followed by sapropterin dihydrochloride and vitamin C
  Treatment Regimen 1: Sapropterin dihydrochloride 5 mg/kg twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14.
  Treatment Regimen 2: Sapropterin dihydrochloride 5 mg/kg + 500 mg vitamin C twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 28
  The washout period of 1 day comprised between treatment regimens.
- Sapropterin Dihydrochloride 10mg/kg and Vitamin C First, Then Sapropterin Dihydrochloride 10mg/kg: Sequence B: Sapropterin dihydrochloride and vitamin C as the first treatment followed by sapropterin dihydrochloride
  Treatment Regimen 2: Sapropterin dihydrochloride 5 mg/kg + 500 mg vitamin C twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14.
  Treatment Regimen 1: Sapropterin dihydrochloride 5 mg/kg twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal Day 28.
  The washout period of 1 day comprised between treatment regimens.
- Total: Total of all reporting groups
Arm/Group | Sapropterin Dihydrochloride 10mg/kg First, Then Sapropterin Dihydrochloride 10mg/kg and Vitamin C | Sapropterin Dihydrochloride 10mg/kg and Vitamin C First, Then Sapropterin Dihydrochloride 10mg/kg | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (12.1) | 43.2 (14.0) | 42.9 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 16 | 16 | 32
Age [Count of Participants; unit: Participants]
  < 65 Years | 24 | 22 | 46
  ≥ 65 Years | 0 | 2 | 2
Race [Count of Participants; unit: Participants]
  White | 10 | 15 | 25
  Black/African American | 13 | 8 | 21
  Other | 1 | 1 | 2
Ethnicity [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 18 | 17 | 35
  Hispanic or Latino | 6 | 7 | 13
Weight [Mean (Standard Deviation); unit: kg] | 95.78 (18.36) | 96.80 (16.93) | 96.29 (17.48)
Height [Mean (Standard Deviation); unit: cm] | 170.81 (8.47) | 172.71 (9.98) | 171.76 (9.21)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.33 (5.62) | 32.45 (5.70) | 32.39 (5.60)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC0-12hrs) of Plasma BH4 Concentration
Description: Plasma BH4 concentration area under the curve (AUC0-12 hrs) at the end of each regimen in subjects with endothelial dysfunction.
Time Frame: At 30 minutes prior to dosing, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0, 10.0, and 12.0 hours after dosing.
Population: Intent-to-treat (ITT) Population
Measure: Mean (Standard Deviation); unit: nM*hr
Groups:
- Sapropterin Dihydrochloride 10 mg/kg: Sapropterin dihydrochloride 5 mg/kg twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14 or Day 28.
- Sapropterin Dihydrochloride+Vitamin C 10 mg/kg: Sapropterin dihydrochloride 5 mg/kg and 500 mg Vitamin C twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14 or Day 28.
Arm/Group | Sapropterin Dihydrochloride 10 mg/kg | Sapropterin Dihydrochloride+Vitamin C 10 mg/kg
Number analyzed (Participants) | 44 | 43
nM*hr | 633 (286) | 993 (545)
Statistical Analysis 1: Comparison: Sapropterin Dihydrochloride 10 mg/kg vs Sapropterin Dihydrochloride+Vitamin C 10 mg/kg; To determine if administration of saproprterin dihydrochloride administered with Vitamin C results in higher plasma BH4 concentrations when compared with administration of sapropterin dihydrochloride alone in subjects with endothelial dysfunction. The difference in the plasma BH4 concentration (AUC0-12 hr) between the 2 regimens will be compared using a mixed model with a 0.05 level of significance. The difference is represented as the geometric mean ratio; Test type: Superiority; p < 0.001, Mixed Models Analysis — The model will constitute the independent variables of treatment regimen, treatment sequence, and period as fixed effects, and subject as a random effect. The dependent variable plasma BH4 concentration (AUC0-12 hr) expressed in log transformation; Geometric Mean Ratio = 1.5, 95% CI 2-sided [1.2 to 1.8]

2. Secondary Outcome: Area Under the Curve (AUC0-12hrs) of Plasma BH2 and B Concentration
Description: Plasma BH2 and B concentration area under the curve (AUC0-12hrs) at the end of each regimen in subjects with endothelial dysfunction.
Time Frame: At 30 minutes prior to dosing, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0, 10.0, and 12.0 hours after dosing.
Population: ITT population
Measure: Mean (Standard Deviation); unit: nM*hr
Groups:
- Sapropterin Dihydrochloride: Sapropterin dihydrochloride 5 mg/kg twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14 or Day 28.
- Sapropterin Dihydrochloride+Vitamin C: Sapropterin dihydrochloride 5 mg/kg and 500 mg Vitamin C twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14 or Day 28.
Arm/Group | Sapropterin Dihydrochloride | Sapropterin Dihydrochloride+Vitamin C
Number analyzed (Participants) | 44 | 43
nM*hr
  BH2 | 875 (455) | 772 (376)
  B | 231 (163) | 185 (123)
Statistical Analysis 1: Comparison: Sapropterin Dihydrochloride vs Sapropterin Dihydrochloride+Vitamin C; To determine if administration of saproprterin dihydrochloride administered with Vitamin C results in higher plasma BH2 when compared with administration of sapropterin dihydrochloride alone in subjects with endothelial dysfunction. The difference in the plasma BH2 concentration (AUC0-12 hr) between the 2 regimens will be compared using a mixed model with a 0.05 level of significance. The difference is represented as the geometric mean ratio; Test type: Superiority; p = 0.139, Mixed Models Analysis — The model will constitute the independent variables of treatment regimen, treatment sequence, and period as fixed effects, and subject as a random effect. The dependent variable plasma BH2 concentration (AUC0-12 hr) expressed in log transformation; Geometric Mean Ratio = 0.9, 95% CI 2-sided [0.7 to 1.0]
Statistical Analysis 2: Comparison: Sapropterin Dihydrochloride vs Sapropterin Dihydrochloride+Vitamin C; To determine if administration of saproprterin dihydrochloride administered with Vitamin C results in Total B (biopterin) when compared with administration of sapropterin dihydrochloride alone in subjects with endothelial dysfunction. The difference in the Total B (biopterin) concentration (AUC0-12 hr) between the 2 regimens will be compared using a mixed model with a 0.05 level of significance. The difference is represented as the geometric mean ratio; Test type: Superiority; p = 0.570, Mixed Models Analysis — The model will constitute independent variables of treatment regimen, treatment sequence, and period as fixed effects, and subject as a random effect. The dependent variable Total B concentration (AUC0-12 hr) expressed in log transformation; Geometric Mean Ratio = 0.96, 95% CI 2-sided [0.83 to 1.11]

3. Secondary Outcome: Area Under the Curve (AUC0-12hours) for Calculated BH4 (From Total Biopterin)
Description: Total biopterin concentration area under the curve (AUC0-12hours) at the end of each regimen in subjects with endothelial dysfunction is theoretically the sum of BH4, BH2 and B. Biopterin is the metabolite of BH4 after oxidative conversion of BH4 and BH2 to biopterin. Total biopterin concentrations represent the summation of drug and metabolites: BH4, BH2 and B. The total biopterin concentrations can be converted to BH4 concentration using the conversion factor 2.150.
Time Frame: At 30 minutes prior to dosing, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0, 10.0, and 12.0 hours after dosing.
Population: ITT population
Measure: Mean (Standard Deviation); unit: nM*hr
Arm/Group | Sapropterin Dihydrochloride | Sapropterin Dihydrochloride+Vitamin C
Number analyzed (Participants) | 44 | 43
nM*hr | 440 (183) | 440 (211)

4. Secondary Outcome: Ratio of BH2, B and BH4 Calculated From Total Biopterin Area Under the Curve (0-12hours) for Subjects Administered Sapropterin Dihydrochloride With Vitamin C to Subjects Administered Sapropterin Alone.
Description: Ratio of Mean AUC (0-12 hours) for subjects receiving (Sapropterin dihydrochloride + Vitamin C)/ Mean AUC (0-12 hours) for subjects receiving Sapropterin dihydrochloride alone) for BH4, BH2, B, BH4/BH2 Ratio, and BH4 Calculated from Total Biopterin.
Time Frame: At 30 minutes prior to dosing, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0, 10.0, and 12.0 hours after dosing.
Population: ITT population. AUC (0 to 12 hour) means were calculated for 44 subjects in the Sapropterin dihydrichloride and 43 subjects on Sapropterin dihydrochloride + Vitamin C
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- (Sapropterin Dihydrochloride+Vitamin C)/(Sapropterin Dihydrochloride): Ratio of Mean AUC (0-12hours) for all subjects (44) receiving sapropterin dihydochloride + Vitamin C/ Mean AUC (0-12 hours) for all subjects (43) receiving sapropterin dihydochloride alone.
Arm/Group | (Sapropterin Dihydrochloride+Vitamin C)/(Sapropterin Dihydrochloride)
Number analyzed (Participants) | 44
ratio
  BH2 | 0.998 (0.577)
  B | 1.04 (1.10)
  Calculated BH4 (from Total Biopterin) | 1.03 (0.33)

5. Secondary Outcome: Change From Baseline in Peripheral Arterial Tonometry (PAT)
Description: PAT measures pulse wave amplitude of the small arteries of the finger as a surrogate to assess endothelial function and arterial stiffness using a finger plethysmographic probe and 5-minute occlusion of the brachial artery. Endothelial dysfunction, a protocol inclusion criteria, is defined by an abnormal PAT of < or = 1.70. Change is calculated as follows: end time measurement - starting time measurement.
Time Frame: At Baseline, Day 13 and Day 27
Population: ITT population.
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Sapropterin Dihydrochloride 10mg/kg: Sapropterin dihydrochloride 5 mg/kg twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14 or Day 28.
  The washout period of 1 day comprised between treatment regimens.
- Sapropterin Dihydrochloride 10mg/kg and Vitamin C: Sapropterin dihydrochloride 5 mg/kg + 500 mg vitamin C twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14 or Day 28
Arm/Group | Sapropterin Dihydrochloride 10mg/kg | Sapropterin Dihydrochloride 10mg/kg and Vitamin C
Number analyzed (Participants) | 44 | 43
Ratio
  Baseline: number analyzed (Participants) | 24 | 24
  Baseline | 1.5113 (0.1669) | 1.4859 (0.1437)
  Day 13: number analyzed (Participants) | 21 | 23
  Day 13 | 1.8509 (0.4677) | 1.7754 (0.3760)
  Change from Baseline to Day 13: number analyzed (Participants) | 21 | 23
  Change from Baseline to Day 13 | 0.3467 (0.4311) | 0.2902 (0.4329)
  Day 27: number analyzed (Participants) | 23 | 20
  Day 27 | 1.9047 (0.4903) | 1.6482 (0.4250)
  Change from Day 13 to Day 27: number analyzed (Participants) | 23 | 20
  Change from Day 13 to Day 27 | 0.1293 (0.4897) | -0.1641 (0.4294)
Statistical Analysis 1: Comparison: Sapropterin Dihydrochloride 10mg/kg vs Sapropterin Dihydrochloride 10mg/kg and Vitamin C; The raw value of PAT obtained from the first period (baseline to Day 13) will be used to compare the two treatments; Test type: Superiority; p = 0.593, ANCOVA; The model will have the treatments and the baseline measurement as independent variables and measurement at Day 13 as the dependent variable

6. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP)
Description: Change is calculated as follows: end time measurement - starting time measurement.
  Mean daytime systolic blood pressure measured by ambulatory blood pressure monitoring (ABPM)
Time Frame: At Baseline, Day 13 and Day 27
Population: ITT population
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Sapropterin dihydrochloride10mg/kg: Sapropterin dihydrochloride 5 mg/kg twice a day administered as whole tablets orally within 1 hour after morning and evening meals and the last dose within 1 hour after a morning meal on Day 14 or Day 28.
Arm/Group | Sapropterin dihydrochloride10mg/kg | Sapropterin Dihydrochloride 10mg/kg and Vitamin C
Number analyzed (Participants) | 23 | 20
mm Hg
  Baseline: number analyzed (Participants) | 16 | 15
  Baseline | 125.14 (13.42) | 131.29 (13.05)
  Change from Baseline to Day 13: number analyzed (Participants) | 9 | 11
  Change from Baseline to Day 13 | -3.24 (8.64) | -0.10 (6.53)
  Change from Day 13 to Day 27: number analyzed (Participants) | 14 | 9
  Change from Day 13 to Day 27 | -1.67 (7.29) | 3.31 (6.43)

7. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP)
Description: Change is calculated as follows: end time measurement - starting time measurement.
  Mean daytime diastolic blood pressure measured by ambulatory blood pressure monitoring (ABPM)
Time Frame: At Baseline, Day 13 and Day 27
Population: ITT population
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Sapropterin dihydrochloride10mg/kg: Sapropterin dihydrochloride 5 mg/kg twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14 or Day 28..
Arm/Group | Sapropterin dihydrochloride10mg/kg | Sapropterin Dihydrochloride 10mg/kg and Vitamin C
Number analyzed (Participants) | 23 | 20
mm Hg
  Baseline: number analyzed (Participants) | 16 | 15
  Baseline | 77.32 (11.05) | 80.15 (14.05)
  Change from Baseline to Day 13: number analyzed (Participants) | 9 | 11
  Change from Baseline to Day 13 | -2.31 (6.84) | 0.45 (5.31)
  Change from Day 13 to Day 27: number analyzed (Participants) | 14 | 9
  Change from Day 13 to Day 27 | -2.01 (6.60) | 1.23 (5.21)

8. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs)
Description: A treatment-emergent Adverse Events (TEAE) is any Adverse Events that newly appeared, increased in frequency or worsened in severity following initiation of study drug administration.
Time Frame: Up to 56 ± 3 Days.
Population: ITT and Safety Population. Four subjects enrolled in the study before changing from a parallel to a cross over study not reflected in the data table in the Participant Flow module. Two subjects received sapropterin dihydrochloride only and two subjects received sapropterin dihydrichloride + vitamin C only.
Measure: Count of Participants; unit: Participants
Arm/Group | Sapropterin Dihydrochloride | Sapropterin Dihydrochloride+Vitamin C
Number analyzed (Participants) | 49 | 50
Participants
  Subjects with any Adverse Event | 19 | 16
  Subjects with any Serious Adverse Event | 0 | 0
  Subjects with any treatment-related Adverse Event | 16 | 13
  Any treatment-related Serious Adverse Event | 0 | 0
  Death | 0 | 0
  Any AEs Leading to Study Discontinuation | 1 | 0

9. Secondary Outcome: Change From Baseline in Urinary 8-isoprostane/Creatinine
Description: Biomarkers of endothelial function, oxidative stress, and inflammation as measured by 8-isoprostane.
Time Frame: At Baseline, Day 14 and Day 28
Population: ITT Population
Measure: Mean (Standard Deviation); unit: pg/mg
Groups:
- Sapropterin Dihydrochloride 10mg/kg: Sapropterin dihydrochloride 5 mg/kg twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14 or Day 28.
- Sapropterin dihydrochloride10mg/kg and Vitamin C: Sapropterin dihydrochloride 5 mg/kg + 500 mg vitamin C twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14 or Day 28..
Arm/Group | Sapropterin Dihydrochloride 10mg/kg | Sapropterin dihydrochloride10mg/kg and Vitamin C
Number analyzed (Participants) | 42 | 41
pg/mg
  Baseline: number analyzed (Participants) | 21 | 23
  Baseline | 898.01 (671.25) | 992.38 (569.80)
  Change from Baseline to Day 14: number analyzed (Participants) | 21 | 21
  Change from Baseline to Day 14 | -192.13 (529.16) | -31.75 (664.40)
  Change from Day 14 to Day 28: number analyzed (Participants) | 21 | 20
  Change from Day 14 to Day 28 | -117.61 (472.61) | 32.44 (364.60)

10. Secondary Outcome: Change From Baseline in Cyclic Guanosine Monophosphate (cGMP)
Description: Biomarkers of endothelial function, oxidative stress, and inflammation as measured by cyclic guanosine monophosphate (cGMP).
Time Frame: At Baseline, Day 14 and Day 28.
Population: ITT Population
Measure: Mean (Standard Deviation); unit: pmol/mL
Groups:
- Sapropterin Dihydrochloride 10mg/kg Vitamin C: Sapropterin dihydrochloride 5 mg/kg twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14 or Day 28.
Arm/Group | Sapropterin Dihydrochloride 10mg/kg Vitamin C | Sapropterin dihydrochloride10mg/kg and Vitamin C
Number analyzed (Participants) | 43 | 42
pmol/mL
  Baseline: number analyzed (Participants) | 21 | 23
  Baseline | 3.7941 (1.1839) | 3.8533 (1.4658)
  Change from Baseline to Day 14: number analyzed (Participants) | 21 | 22
  Change from Baseline to Day 14 | 0.6278 (2.0258) | 0.2088 (1.3248)
  Change from Day 14 to Day 28: number analyzed (Participants) | 22 | 20
  Change from Day 14 to Day 28 | -0.0507 (1.1369) | -0.0078 (1.9556)

11. Secondary Outcome: Change in Urinary Albumin to Creatinine Ratio (mg/g)
Description: Change in Urinary Albumin to Creatinine Ratio (mg/g) from Baseline to Day 14, Baseline to Day 28, and from Day 14 to Day 28
Time Frame: Baseline, Day 14 and Day 28
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Sapropterin Dihydrochloride 10mg/kg | Sapropterin Dihydrochloride 10mg/kg and Vitamin C
Number analyzed (Participants) | 20 | 21
mg/g
  Baseline: number analyzed (Participants) | 14 | 18
  Baseline | 13.3 (35.7) | 12.3 (19.0)
  Change from Baseline to Day 14: number analyzed (Participants) | 10 | 12
  Change from Baseline to Day 14 | -1.2 (17.9) | 2.7 (18.6)
  Change from Day 14 to Day 28: number analyzed (Participants) | 10 | 9
  Change from Day 14 to Day 28 | -2.2 (4.9) | 4.9 (10.2)

12. Secondary Outcome: Number of Participants With Urinary Albumin to Creatinine Ratio <30 mg/g
Description: Summary of Urinary Albumin to Creatinine Ratio (mg/g) by subjects with ratio <30 mg/g and subjects with ratios >=30 mg/g at Baseline, Day 14 and Day 28
Time Frame: Baseline, Day 14 and Day 28
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Sapropterin Dihydrochloride 10mg/kg | Sapropterin Dihydrochloride 10mg/kg and Vitamin C
Number analyzed (Participants) | 27 | 30
Participants
  Baseline < 30 mg/g: number analyzed (Participants) | 14 | 18
  Baseline < 30 mg/g | 13 | 16
  Baseline >=30 mg/g: number analyzed (Participants) | 14 | 18
  Baseline >=30 mg/g | 1 | 2
  Day 14 < 30 mg/g: number analyzed (Participants) | 12 | 14
  Day 14 < 30 mg/g | 10 | 13
  Day 14 >=30 mg/g: number analyzed (Participants) | 12 | 14
  Day 14 >=30 mg/g | 2 | 1
  Day 28 < 30 mg/g: number analyzed (Participants) | 13 | 12
  Day 28 < 30 mg/g | 12 | 10
  Day 28 >=30 mg/g: number analyzed (Participants) | 13 | 12
  Day 28 >=30 mg/g | 1 | 2

ADVERSE EVENTS:
Time Frame: Up to 56 ± 3 Days.
Description: Four subjects enrolled in the study before changing from a parallel to a cross over study and therefore are not reflected in the data table in the Participant Flow module. Two subjects received sapropterin dihydrochloride only and two subjects received sapropterin dihydrochloride + vitamin C only.
Groups:
- Sapropterin Dihydrochloride 10mg/kg: Sapropterin dihydrochloride 5 mg/kg twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14.
  The washout period of 1 day comprised between treatment regimens.
- Sapropterin Dihydrochloride 10mg/kg and Vitamin C: Sapropterin dihydrochloride 5 mg/kg + 500 mg vitamin C twice a day administered as whole tablets orally within 1 hour after morning and evening meals for 13 days and the last dose within 1 hour after a morning meal on Day 14.
  The washout period of 1 day comprised between treatment regimens.
Arm/Group | Sapropterin Dihydrochloride 10mg/kg | Sapropterin Dihydrochloride 10mg/kg and Vitamin C
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 19/49 | 16/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sapropterin Dihydrochloride 10mg/kg (N=49) | Sapropterin Dihydrochloride 10mg/kg and Vitamin C (N=50)
Diarrhoea (Gastrointestinal disorders) | 5 | 5
Stomach discomfort (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Headache (Nervous system disorders) | 4 | 4
Dysgeusia (Nervous system disorders) | 1 | 0
Thirst (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 0
Pharmaceutical product complaint (General disorders) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 2
Blood lactate dehydrogenase abnormal (Investigations) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Intertrigo candida (Infections and infestations) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days